CLINICAL TRIAL: NCT05928494
Title: The Effect of Scenario Based High Reality Simulation Method on Problem Solving Skills and Anxiety Levels of Midwifery Students
Brief Title: The Effect of High Reality Simulation Method on Problem Solving Skills and Anxiety Levels of Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBÜ-AYDINKARTAL-003
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Care
Keywords: Problem Solving Skill; Simulation; Midwifery; State Anxiety; Student
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (n:39) (Experimental): Postpartum care applications were carried out with the high-reality Gaumard Scientific brand, product code: S550.100 Noella simulator in the simulation laboratory of the midwifery department to the students in the intervention group.
  Interventions: Other: Scenario-based high-fidelity simulation method
- Control group (n:39) (No Intervention): Postpartum care practices were performed on the standard adult patient model in the basic skills laboratory of the midwifery department for the students in the control group.

INTERVENTIONS:
Other: Scenario-based high-fidelity simulation method — Postpartum care applications were carried out with the high-reality Gaumard Scientific brand, product code: S550.100 Noella simulator in the simulation laboratory of the midwifery department to the students in the intervention group.
  Arms: İntervention group (n:39)

SUMMARY:
This study was planned to determine the effect of scenario-based high-fidelity simulation method on the application problem solving skills and anxiety levels of the 3rd year students of Health Sciences University Hamidiye Health Sciences Faculty Midwifery Department. The research, which is planned in a experimental design, will be carried out with Istanbul Health Sciences University Hamidiye Health Sciences Faculty 3rd year midwifery (N:80) students. Students participating in the study will be divided into intervention (n:40) and control (n:40) groups according to the computer-assisted simple random sampling technique. Intervention group students will be given an application about postpartum care on a standard adult patient model in the high-validity simulation laboratory accompanied by a scenario, and control group students will be made in the vocational skills laboratory. "Descriptive Information Form", "State Anxiety Inventory", "Problem Solving Inventory" and "Satisfaction Questionnaire with Educational Methods" will be applied to the students participating in the research.

DETAILED DESCRIPTION:
This study was planned to determine the effect of scenario-based high-fidelity simulation method on the application problem solving skills and anxiety levels of the 3rd year students of Health Sciences University Hamidiye Health Sciences Faculty Midwifery Department.

The universe of the research consisted of 3rd grade students who took the "Risky Birth and Postpartum Period" course in the Midwifery Department of the Faculty of Health Sciences of Hamidiye in the spring semester of the 2021-2022 academic year (N:80). Students who volunteered to participate in the study were included in the study. Computer-assisted randomization will be used in the study, and random assignment was made to the intervention (n:40) and control (n:40) groups by entering the number of cases through the program with the URL address https://www.randomizer.org. Before the application, the "Informed Voluntary Consent Form" was shared with the students and their consent was obtained.

All groups were informed before the applications. In this context, a question-and-answer session was held by giving information about the applications to be made regarding the research. The students were given information about the introduction of the simulator and the model, the flow chart of the training plan, the content of the training plan, the environment, the locations of the materials. Before the application, all groups were given theoretical information about postpartum care for 2 hours with a power point presentation. After the information, the "Descriptive Information Form" was applied to the students, and the "State Anxiety Inventory" and "Problem Solving Inventory" were applied as a pre-test. Postpartum care applications were carried out for the students in the intervention group on a high-reality Gaumard Scientific brand, product code: S550.100 Noella simulator in the simulation laboratory of the Midwifery department, and on the standard adult patient model in the basic skills laboratory for the control group students. After the training, "State Anxiety Inventory", "Problem Solving Inventory" and "Satisfaction Questionnaire with Educational Methods" were applied to all students as a post-test.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research.
* Being a third year student at SBU, Hamidiye Faculty of Health Sciences, Midwifery Department.
* To have successfully completed the theory and practice of basic principles and practices in midwifery.
* To have taken the risky birth and postpartum period lesson.

Exclusion Criteria:

* Not volunteering to participate in the research.
* Not to be a third year student at the Faculty of Health Sciences, Hamidiye, Department of Midwifery.
* Not having successfully completed the theory and practice of basic principles and practices in midwifery.
* Not having taken the risky birth and postpartum lesson.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  In this form, which was created by the researchers based on the literature, the participants' age, the high school they graduated from, the education level of their parents, their willingness to choose the profession, their feeling of belonging to the profession, etc. questions are included.
State Anxiety Inventory | 10 minutes
  The scale consists of two subscales, continuous and state, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how the individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how the individual feels independently of the situation and conditions. The scores obtained from the scale theoretically vary between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
Problem Solving Inventory | 10 minutes
  Originally, the problem solving inventory was applied to prospective teachers by Heppner and Petersen, and the Cronbach Alpha internal consistency coefficient obtained for all of them was found to be 0.90. Erenler applied the inventory to nurses and found the Cronbach Alpha coefficient to be 0.77. These results show that the inventory is valid and reliable. However, in the literature, it is seen that the problem solving inventory is also used in studies in the field of nursing. In the problem solving inventory, each question is given a score between 1 and 6. In the scoring of the inventory, the lowest score is 32 and the highest score is 192. The high total scores obtained from the scale are interpreted that the individual perceives himself/herself as inadequate in problem solving skills.

SECONDARY OUTCOMES:
State Anxiety Inventory | 10 minutes
  The scale consists of two subscales, continuous and state, each consisting of 20 questions. It can be applied to individuals over the age of 14. The state anxiety scale determines how the individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how the individual feels independently of the situation and conditions. The scores obtained from the scale theoretically vary between 20 and 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
Problem Solving Inventory | 10 minutes
  Originally, the problem solving inventory was applied to prospective teachers by Heppner and Petersen, and the Cronbach Alpha internal consistency coefficient obtained for all of them was found to be 0.90. Erenler applied the inventory to nurses and found the Cronbach Alpha coefficient to be 0.77. These results show that the inventory is valid and reliable. However, in the literature, it is seen that the problem solving inventory is also used in studies in the field of nursing. In the problem solving inventory, each question is given a score between 1 and 6. In the scoring of the inventory, the lowest score is 32 and the highest score is 192. The high total scores obtained from the scale are interpreted that the individual perceives himself/herself as inadequate in problem solving skills.
Satisfaction Survey with Training Methods | 10 minutes
  The questionnaire consists of 16 propositions. One of these propositions is the proposition "I am satisfied with this education method in general", which questions the state of being satisfied with the education. Other propositions were formed from propositions aiming to determine the views of the education method in general about the contribution of the education method to the learning and professional life of the student. Each proposition is scored on a 5-point Likert scale (1-strongly disagree, 5-strongly agree). It is determined that as the scale score average increases, students' satisfaction with the education method increases, and as the scale score average decreases, their satisfaction with the education method decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin AYDIN KARTAL Assoc. Prof. Dr., Principal Investigator — Saglik Bilimleri Universitesi; Sema AKER Research Assıstant, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No